CLINICAL TRIAL: NCT03119506
Title: Effects of Recess Timing and Activity on Children's Eating Behaviors
Status: Completed | Type: Observational
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Naiman Khan, Assistant Professor, University of Illinois at Urbana-Champaign
Other Study IDs: 16379
Record Dates: First submitted 2017-04-10; First posted 2017-04-18 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Physical Activity; Diet Habit; Health Behavior
MeSH Terms: conditions — Motor Activity; Feeding Behavior; Health Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Long Recess Duration/Before Lunch
  Interventions: Behavioral: Recess
- Short Recess Duration/Before Lunch
  Interventions: Behavioral: Recess
- Long Recess Duration/After Lunch
  Interventions: Behavioral: Recess
- Short Recess Duration/After Lunch
  Interventions: Behavioral: Recess

INTERVENTIONS:
Behavioral: Recess — Recess timing and duration effects on lunch intake

SUMMARY:
This study aims to understand the interaction between school recess activity and duration and lunch choices among elementary school children

ELIGIBILITY:
Inclusion Criteria:

* Parental/guardian consent
* 8-11 years of age

Exclusion Criteria:

* No parental/guardian consent
* Below 8 years and above 11 years

Ages: 8 Years to 11 Years | Sex: All
Age Groups: Child
Study Population: Elementary School Children
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-02-27 (Actual)

PRIMARY OUTCOMES:
Objectively Measured Physical Activity during Recess | Immediately following or before lunch

SECONDARY OUTCOMES:
Executive Function | Measured within 1 week of Physical Activity Assessment
  Early Adolescent Temperament and Trail Making Questionnaire
Weight Status | Measured within 1 week of Physical Activity Assessment
Plate Waste at Lunch | Immediately following or before recess